CLINICAL TRIAL: NCT01920373
Title: Platelet-Rich Plasma Versus Corticosteroid Injection as Treatment for Degenerative Pathology of the Temporomandibular Joint
Brief Title: Platelet-Rich Plasma vs Corticosteroid Injection as Treatment for Degenerative Pathology of the Temporomandibular Joint
Status: Withdrawn | Phase: Phase 1 | Type: Interventional
Why Stopped: The study was cancelled.
Sponsor: Kaiser Permanente (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: 468485
Record Dates: First submitted 2013-08-08; First posted 2013-08-12 (Estimated); Last update posted 2015-03-11 (Estimated); Status verified 2015-03

CONDITIONS: Degenerative Joint Disease
Keywords: degenerative joint disease; temporomandibular joint
MeSH Terms: conditions — Joint Diseases

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Group A (corticosteroid injection group) (Active Comparator): Group A will receive one intra-articular injection of 2 ml of solution containing 1ml of 10mg/ml Triamcinolone suspended in 1 ml of 0.5% Bupivacaine solution per affected joint
  Interventions: Drug: Group A (corticosteroid injection group)
- Group B (platelet rich plasma injection) (Experimental): Group B will receive a 2 ml intra-articular injection of a platelet rich plasma preparation per affected joint
  Interventions: Biological: Group B (platelet rich plasma injection group)

INTERVENTIONS:
Drug: Group A (corticosteroid injection group)
  Arms: Group A (corticosteroid injection group)
Biological: Group B (platelet rich plasma injection group)
  Arms: Group B (platelet rich plasma injection)

SUMMARY:
1.0 BACKGROUND AND HYPOTHESES

1.1 Osteoarthritis is a continuous and entirely physiologic adaptive process that occurs in every joint. These include the replication of cells that produce matrix, enzymes, protease inhibitors, cytokines, and other peptides. Along with the synthesis of new tissue there is a release of breakdown products into the synovial fluid. Enzymes and phagocytes are required to clear these breakdown products. Normal tissue turnover involves synthesis and breakdown in well-regulated balance. In the degenerative state this balance is upset producing inflammation-derived alterations to the synovium, cartilage, capsule, tendons, and bone. Common causes of such alterations include increased loading, physical stress, and traumatic injury to the joint.

1.2 The rationale for the use of corticosteroids in temporomandibular joint therapy is that they inhibit prostaglandin synthesis and decrease the activity of collagenase and other enzymes that degrade the articular cartilage. Platelet rich plasma is a novel therapeutic agent that has several potential advantages over corticosteroids for the treatment of degenerative pathology of the temporomandibular joint. Platelet rich plasma has been shown to have anti-inflammatory, analgesic, and anti-bacterial properties. It also restores intra-articular hyaluronic acid, increases glycosaminoglycan condrocyte synthesis, balances joint angiogenesis, and provides a scaffold for stem cell migration. Autologous platelet rich plasma injections for treatment of knee cartilage degenerative lesions and osteoarthritis have shown longer efficacy than hyaluronic acid injections in reducing pain and recovering articular function. Similarly, platelet rich plasma has shown to have better outcomes than corticosteroid injections in the management of lateral epicondylitis, and better outcomes than hyaluronic acid injections in the management of osteochondral lesions of the talus.

1.3 Current treatments for degeneration and osteoarthritis of the temporomandibular joint are focused primarily on palliation by reducing inflammation and inflammatory mediators. This study seeks to validate a therapeutic agent that has the potential to actively prevent the progression of degeneration in addition to reducing pain and inflammation

DETAILED DESCRIPTION:
2.0 OBJECTIVES AND PURPOSE

2.1 The purpose of this study is to compare the efficacy, in terms of pain relief and improvement in function, of intra-articular injections with platelet rich plasma versus the current standard which is corticosteroid injections into the temporomandibular joint.

ELIGIBILITY:
Inclusion Criteria: The following diagnostic criteria for patient selection are to be used:

* Patients will need to have a history of chronic pain (at least 3 months) refractory to conservative therapy with non-steroidal anti-inflammatory medications, muscle relaxants, diet modifications and splint therapy
* Patients will also need to have imaging findings (radiography or magnetic resonance imaging) that show mild to severe degenerative changes of the temporomandibular joint

Exclusion Criteria: Exclusion criteria will include

* Patients with systemic disorders such as rheumatic diseases, hematologic diseases, active infections, immunosuppression
* Patients receiving therapy with anticoagulants

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2013-11; Primary Completion 2013-11 (Actual)

PRIMARY OUTCOMES:
Pain relief | 24 weeks
  Changes in pain relief will be evaluated at 1, 3, and six month intervals using the Pain resource centers TMJ scale.

SECONDARY OUTCOMES:
Improvement in function | 24 weeks
  The patients improvement in function will be evaluated at 1,3, and 6 months for improvement using the pain resource centers TMJ scale.

CONTACTS AND LOCATIONS:
Overall Officials: Husam G Elias, MD, DMD, Principal Investigator — Kaiser Permanente; Julian J Wilson, DDS, Study Chair — Kaiser Permanente
Locations (1):
- Kaiser Permanente Los Angeles Medical Center, Los Angeles, California, United States